CLINICAL TRIAL: NCT07366060
Title: Evaluation of the Effectiveness of Third Occipital Nerve Pulsed Radiofrequency Treatment in Patients With Cervicogenic Headache
Brief Title: Effectiveness of Third Occipital Nerve Pulsed Radiofrequency in Cervicogenic Headache
Acronym: TON-PRF-CH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hatice Babaoğlan, medical doctor, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TABED 1-25-1390
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cervicogenic Headache; Third Occipital Nerve
Keywords: cervicogenic headache; Pulsed Radiofrequency; Third Occipital Nerve; TON PRF
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: All participants will receive ultrasound-guided third occipital nerve pulsed radiofrequency treatment, and outcomes will be compared with baseline measurements during follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TON PRF Treatment (Experimental): Participants diagnosed with cervicogenic headache who demonstrate a positive response to diagnostic third occipital nerve block will receive ultrasound-guided pulsed radiofrequency treatment of the third occipital nerve.
  Interventions: Procedure: Third Occipital Nerve Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Third Occipital Nerve Pulsed Radiofrequency — Ultrasound-guided pulsed radiofrequency treatment applied to the third occipital nerve at the C2-3 zygapophyseal joint level for the management of cervicogenic headache.

SUMMARY:
Cervicogenic headache is a secondary headache disorder originating from cervical spine structures and is frequently associated with chronic pain, functional limitation, and impaired quality of life. The third occipital nerve, which innervates the C2-3 zygapophyseal joint, plays an important role in the pathophysiology of cervicogenic headache.

Pulsed radiofrequency is a minimally invasive interventional pain management technique that modulates nociceptive transmission without causing permanent neural damage. Although third occipital nerve pulsed radiofrequency is increasingly used in clinical practice, prospective data evaluating its clinical effectiveness and safety remain limited.

The aim of this prospective, single-center study is to evaluate the effectiveness and safety of ultrasound-guided third occipital nerve pulsed radiofrequency treatment in patients diagnosed with cervicogenic headache. Pain intensity, headache characteristics, analgesic consumption, and patient-reported outcomes will be assessed before treatment and during follow-up. The results of this study are expected to contribute to clinical evidence supporting interventional treatment strategies for cervicogenic headache.

DETAILED DESCRIPTION:
Cervicogenic headache is a chronic secondary headache disorder arising from cervical spine structures, particularly the C2-3 zygapophyseal joint and its innervating third occipital nerve. This condition is often resistant to conservative therapies and may significantly impair daily functioning and sleep quality.

Pulsed radiofrequency is a neuromodulatory technique that delivers intermittent high-frequency electrical current while maintaining tissue temperatures below neurodestructive thresholds. This approach is believed to reduce pain by altering nociceptive signal transmission and inflammatory processes without causing permanent nerve injury.

This study is designed as a prospective, single-center, open-label, interventional clinical study conducted at the Algology Clinic of Ankara City Hospital Bilkent. Adult patients aged 18 years and older who are diagnosed with cervicogenic headache according to the International Classification of Headache Disorders (ICHD-3) criteria and who demonstrate a positive response to ultrasound-guided diagnostic third occipital nerve block will be included.

Eligible patients will undergo ultrasound-guided pulsed radiofrequency treatment of the third occipital nerve at the C2-3 zygapophyseal joint level using standard clinical protocols. Pain intensity will be evaluated using the Visual Analog Scale before the procedure and during follow-up visits at predefined time points. Additional outcome measures will include headache frequency, number of headache days, analgesic medication consumption, impact on daily activities and sleep, and patient-reported global perceived effect.

Follow-up assessments will be conducted at 1, 2, and 3 months after the procedure. All adverse events, complications, and safety-related outcomes associated with diagnostic nerve block and pulsed radiofrequency treatment will be recorded throughout the study period.

The primary objective of this study is to evaluate changes in pain intensity following third occipital nerve pulsed radiofrequency treatment. Secondary objectives include assessment of headache-related disability, medication use, patient satisfaction, and safety outcomes. The findings of this study are expected to provide prospective clinical evidence regarding the effectiveness and safety of third occipital nerve pulsed radiofrequency treatment in patients with cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of cervicogenic headache according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)
* Availability of cranial and cervical spine imaging
* At least 5 headache days per month
* Inadequate response to pharmacological and/or physical therapy treatments
* Ability to understand and provide written informed consent
* Positive response to ultrasound-guided diagnostic third occipital nerve block, defined as at least 50% reduction in pain intensity or patient-reported meaningful improvement

Exclusion Criteria:

* Secondary headache disorders other than cervicogenic headache according to ICHD-3
* Signs or symptoms of cervical nerve root irritation and/or spinal stenosis
* Sensory deficit in the greater occipital nerve dermatome
* Cranio-cervical structural defects or anatomical abnormalities at or near the target site
* Local or systemic infection
* Non-pharmacological headache treatment within the last 3 months (e.g., physical therapy, botulinum toxin A, acupuncture, ozone therapy, cognitive behavioral therapy)
* Pregnancy or suspected pregnancy
* Known allergy to local anesthetic agents
* History of malignancy
* Known organic disease of the brain or spinal cord
* History of cranial or cervical surgery within the last 12 months
* Bleeding or coagulation disorders or use of oral anticoagulant therapy
* Comorbid conditions that may cause headache (e.g., uncontrolled hypertension, intracranial lesions)
* Conditions that may interfere with treatment adherence or outcome assessment (e.g., psychiatric disorders, dementia)
* Request for re-treatment due to development of contralateral pain or other pain conditions during follow-up
* Refusal to undergo the intervention or withdrawal of consent at any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by Visual Analog Scale (VAS) | Baseline, and 1, 2, and 3 months after the procedure
  Pain intensity will be assessed using the Visual Analog Scale (VAS) to evaluate changes in headache-related pain following third occipital nerve pulsed radiofrequency treatment.

SECONDARY OUTCOMES:
Number of headache days per month | Baseline, and 1, 2, and 3 months after the procedure
  The number of days with headache per month will be recorded using patient headache diaries during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim ED, Kim YH, Park CM, Kwak JA, Moon DE. Ultrasound-guided Pulsed Radiofrequency of the Third Occipital Nerve. Korean J Pain. 2013 Apr;26(2):186-90. doi: 10.3344/kjp.2013.26.2.186. Epub 2013 Apr 3. PMID 23614084
- [Result] Lord SM, Barnsley L, Wallis BJ, Bogduk N. Third occipital nerve headache: a prevalence study. J Neurol Neurosurg Psychiatry. 1994 Oct;57(10):1187-90. doi: 10.1136/jnnp.57.10.1187. PMID 7931379
- [Result] Bogduk N. The clinical anatomy of the cervical dorsal rami. Spine (Phila Pa 1976). 1982 Jul-Aug;7(4):319-30. doi: 10.1097/00007632-198207000-00001. PMID 7135065